CLINICAL TRIAL: NCT06589817
Title: A Phase 3, Multicenter, Randomized, Double-blind Study to Evaluate the Efficacy and Safety of Hydrochloride Carliprazine Capsules or Aripiprazole Tablets for the Treatment of Acute Schizophrenia Subjects
Brief Title: A Double-Blind, Randomized Comparative Study of Carliprazine and Aripiprazole in Patients with Acute Schizophrenia
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chengdu Kanghong Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KH734-60101
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Acute Schizophrenia
MeSH Terms: interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hydrochloride Carliprazine capsules + Aripiprazole tablet placebo (Experimental)
  Interventions: Drug: Hydrochloride Carliprazine capsules
- Aripiprazole tablets + Hydrochloride Carliprazine capsules placebo (Active Comparator)
  Interventions: Drug: Aripiprazole tablets

INTERVENTIONS:
Drug: Hydrochloride Carliprazine capsules — Oral administration, once daily, with a total treatment duration of 6 weeks after successful screening.
  Arms: Hydrochloride Carliprazine capsules + Aripiprazole tablet placebo
Drug: Aripiprazole tablets — Oral administration, once daily, with a total treatment duration of 6 weeks after successful screening.
  Arms: Aripiprazole tablets + Hydrochloride Carliprazine capsules placebo

SUMMARY:
This is a non-Inferiority trial to evaluate efficacy and safety of hydrochloride carliprazine capsules and aripiprazole tablets in treating acute schizophrenia in Chinese adults. 376 patients will be randomizdely assigned in a 1:1 ratio to treatment group and control group. All enrolled subjects will be orally administered with hydrochloride carliprazine capsules or aripiprazole tablets for 6 consecutive weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects between 18 and 65 years, male and female;
2. Subjects diagnosed with schizophrenia (according to the DSM-IV criteria);
3. Subjects with a PANSS Total score between 70-120, with a score of at least 4 on two or more of the items of delusions, hallucinatory behavior, conceptual disorganization, or suspiciousness;
4. Subjects with a CGI-S score ≥4;
5. Subjects with a Body Mass Index (BMI) of between 18-40 kg/m2;
6. Subjects and subject's legal guardian or legally acceptable representative have the ability to understand the nature of the trial, agree to comply with the prescribed medication and dosage regimens, complete the scheduled visits, report the adverse events and concomitant medication to investigators, and to be reliably rated on psychiatrically scales，and to provide written informed consent form by subjects and subject's legal guardian or legally acceptable representative.

Exclusion Criteria:

1. Other mental illnesses that meet DSM-5 criteria, excluding schizophrenia, including but not limited to: major depressive disorder, bipolar disorder and related disorders, panic disorder, agoraphobia, social anxiety disorder, obsessive-compulsive disorder, post-traumatic stress disorder, generalized anxiety disorder, bulimia nervosa/anorexia nervosa, neurodevelopmental disorders, schizoaffective disorder, and any other mental illness that may affect subject compliance;
2. Subjects who have been hospitalized for > 21 days for the current acute episode.
3. Subjects with a history of substance abuse or dependence (excluding nicotine or caffeine) in the past 3 months, or those who test positive in the urine drug screening during the screening period (Subjects who test positive in the urine drug screening may be allowed to participate in the study at the researcher's discretion, or may participate if they cease using such substances prior to the trial). Use of narcotic analgesics for a maximum of 3 days is permitted during the trial for clinical medical needs;
4. Subjects who have history of substance abuse or dependence within 3 months, but excluding caffeine and nicotine. Invesgtigators have the right to decide whether subjects who are positive in urine drug screening can be enrolled in the study, or those who have stopped drug use before screening can be enrolled. During the study, the use of up to 3 days of anesthetic analgesics is allowed for medical purposes.
5. Subjects with schizophrenia who are considered resistant/refractory to antipsychotic treatment by history of failure to respond to 2 adequate different antipsychotic medications with a minimum of 6 weeks at clinically efficacious tolerated doses.
6. Subjects who have used long-acting antipsychotic drugs (such as risperidone long-acting injection, paliperidone long-acting injection , fluphenazine, aripiprazole long-acting injection , etc.) within 6 months before screening, or subjects who have received ≥15mg aripiprazole treatment within 14 days before screening.
7. Subjects who have taken >200 mg/day clozapine for any reason, or ≤200 clozapine for the reason other than insomnia, agitation, or anxiety.
8. Subjects with a history of psychosurgerytherapy, electroconvulsive therapy (ECT) or repetitive transcranial magnetic stimulation (rTMS) within 3 months before screening, or those who cannot stop physical therapy during the study.
9. As judged by the investigator, subjects with risk of severe agitation, violent or destructive behaviors (harming self or othres, suicide).
10. Subjects with risk for suicidal behavior during the study as determined by the investigator's clinical assessment and Columbia-Suicide Severity Rating Scale (C-SSRS).
11. Females who are pregnant or breastfeeding, or those are not willing or cannot practice contraceptive methods from the time of signing the ICF to 30 days after the last dose.
12. Subjects with comorbidities that, in the view of the investigator, may interfere with the implementation of the trial or confound the trial results.
13. Subjects with a history of ischemic heart disease or myocardial infarction, congestive heart failure (whether controlled or uncontrolled), angioplasty, stenting, or coronary artery bypass surgery.
14. Subjects with history of central nervous system diesease, including but not limited to stroke, tumor of central nervous system, Parkinson's disease, organic brain disorders, epilepsy or seizures, chronic infections, neurosyphilis, or previously suffered from traumatic brain injury.
15. Subjects with history or presence of clinically significant organic disease, including but not limited to hepatic, renal, pulmonary, cardiovascular, endocrine, neurologic, hematologic, or autoimmunologic diseases.
16. Subjects with history of ophthalmic disease, such as cataract, intraocular surgery (not including corneal refractive surgery), fundus laser therapy, open-angle or angle-closure glaucoma, retinal or corneal disease, severe ocular trauma or its complications, and acute bacterial or viral eye infections within 1 week before screening.
17. Subjects with type I diabetes dellitus or uncontrolled type II diabetes mellitus. Subjects with type II diabetes may be eligible for the trial if their condition is stable as determined by satisfying ALL of the following criteria:

    * HbA1c < 7.0%, and fasting glucose must be ≤ 7.0 mmol/L or non-fasting glucose must be ≤ 11.1 mmol/L at screening, AND
    * If the non-fasting glucose is >11.1mmol/L, subjects must be retested in a fasted state and the retest value must be ≤ 7.0 mmol/L, AND
    * Subjects have maintained a stable regimen of oral anti-diabetic medication(s) for at least 28 days before screening or diabetes has been well-controlled by diet for at least 28 days before screening, AND
    * Subjects have not had any hospitalizations within the 2 months before screening due to diabetes or complications related to diabetes, AND
    * Subjects whose diabetes is not newly diagnosed during screening for the trial.
18. Abnormal hepatic and renal function at screening, sucha as ALT, AST>2×ULN or Cr > 1.2 ×ULN.

(18)Clinically significant abnormal finding on ECG at screening, such as QTcF≥450 ms (male) or ≥470 ms (female).

(19)Positive test for HBsAg, HIV antibody, HCV antibody, and TP-Ab at screening.

(20)If other significant abnormalities in laboratory findings and scales at screening, in the opinion of the investigator, subject is unsuitable for enrollment in the study.

(21)Subjects with uncontrolled hypertension, symptomatic hypotension or orthostatic hypotension.

(22)Subjects with history or presence of tardive dyskinesia or neuroleptic malignant syndrome.

(23)Subjects with history of known allergy to carliprazine capsules, aripiprazole tablets, or their excipients, or highly sensitive person (defined as allergies to more than 2 substances); (24)Subject is unsuitable for enrollment in the study in the opinion of the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
PANSS | week 6
  Change in the Positive and Negative Syndrome Scale (PANSS) score from baseline.

SECONDARY OUTCOMES:
PANSS | week 1.;week 2.;week 4
  Change in the Positive and Negative Syndrome Scale (PANSS) score from baseline.
CGI-S | week 1.;week 2.;week 4.;week 6.
  Change in Clinical Global Impression Severity Scale (CGI-S) score from baseline.
CGI-I | week 1.;week 2.;week 4.;week 6.
  Change in Clinical Global Impression Improvement Scale (CGI-I) score from baseline.
PSP | week 6.
  Change in Personal and Social Performance Scale (PSP) score from baseline.